CLINICAL TRIAL: NCT03214003
Title: Twice-daily Radiotherapy by Simultaneous Integrated Boosting Technique Versus Twice-daily Standard Radiotherapy for Patients With Limited-stage Small Cell Lung Cancer: a Multicenter, Randomized, Controlled, Phase III Study
Brief Title: Twice-daily SIB Radiotherapy Versus Standard Radiotherapy for Patients With SCLC
Acronym: TRISS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Shi, MD (Other)
Collaborators: Sun Yat-sen University (Other); Fudan University (Other); Xijing Hospital (Other); Henan Cancer Hospital (Other Government); Jilin Provincial Tumor Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Air Force General Hospital of the PLA (Other Government); China-Japan Friendship Hospital (Other); Peking University Third Hospital (Other); Peking Union Medical College Hospital (Other); Beijing Hospital (Other Government); Beijing Chao Yang Hospital (Other); Peking University People's Hospital (Other); Peking University First Hospital (Other)
Responsible Party: Sponsor-Investigator, Anhui Shi, MD, associate chief physician, Peking University Cancer Hospital & Institute
Organization: Peking University Cancer Hospital & Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017YJZ19
Record Dates: First submitted 2017-07-05; First posted 2017-07-11 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Small Cell Lung Cancer Limited Stage; Radiotherapy
Keywords: small cell lung cancer limited stage; twice-daily radiotherapy; simultaneous integrated boosting technique
MeSH Terms: interventions — Drug Therapy; Etoposide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIB group (Experimental): Patients in this group will receive concurrent twice-daily radiotherapy by SIB technique (95%PGTV 54Gy, 95%PTV 45Gy,both in 30 twice-daily fractions over 3 weeks, 5 days per week) and chemotherapy (etoposide and cisplatin).
  Interventions: Radiation: SIB
- BID group (Active Comparator): Patients in this group will receive concurrent twice-daily standard radiotherapy (95%PTV 45Gy in 30 twice-daily fractions over 3 weeks, 5 days per week, without SIB) and chemotherapy (etoposide and cisplatin).
  Interventions: Radiation: Standard

INTERVENTIONS:
Radiation: SIB — patients will recieve twice-daily radiotherapy by simultaneous integrated boosting technique concurrent with chemotherapy
  Other Names: chemotherapy with etoposide and cisplatin
  Arms: SIB group
Radiation: Standard — patients will recieve standard twice-daily radiotherapy concurrent with chemotherapy
  Other Names: chemotherapy with etoposide and cisplatin
  Arms: BID group

SUMMARY:
This trial is a multicenter, perspective, non-blinded, randomized controlled phase 3 trial. In order to establish whether the SIB technique can improve the results of twice-daily chemo-RT for patients with LS-SCLC, the investigators will primarily compare survival of patients treated with standard chemotherapy (cisplatin and etoposide) and either SIB twice-daily RT or standard dose twice-daily RT.

DETAILED DESCRIPTION:
Three hundred and twenty-six patients with a histological or cytological proven diagnosis of SCLC will be recruited from 35 centers in 14 areas including provinces, municipalities and autonomous region, from May 2017 to May 2020.

ELIGIBILITY:
Inclusion Criteria:

* Read the patient information and Sign the informed consent before enrollment
* Either sex, age ≥18 and ≤70
* Histologically or cytologically confirmed SLCL
* Limited stage disease(AJCC, 2009 version 7), stage I-III(T any, N any, M0) that can be safely treated with definitive radiation doses, excludes T3-4 due to multiple lung nodules that are too extensive or have tumor/nodal volume that is too large to be encompassed in a tolerable radiation plan, clinical nonmalignant diagnosis by investigator when the pleural is too few to obtain cytological evidence.
* measurable lesion according RECIST 1.1
* PS ECOG 0-1
* having zero to two cycles of systemic chemotherapy with etoposide and cisplatin (cisplatin 60-80 mg/m2 at day1 or divided into two to three days, etoposide 100-120 mg/m2 at day 1 to 3, Q21d, and the treatment delay between two cycles shouldn't be more than 14days).
* patients especially female patients must satisfy the investigator that they are not pregnant, or are not of childbearing potential, or are using adequate contraception. Man must also use adequate contraception
* adequate haematological function: white blood cell ≥3.0×109/L , neutrophils ≥1.5×109/L, platelet ≥100×109/L, hemoglobin ≥90g/L.
* adequate liver and renal function: total bilirubin ≤1.5 ×upper limit normal , alanine transaminase and aspartate aminotransferase ≤1.5 ×upper limit normal, normal serum creatinine and/or calculated creatinine clearance ≥60ml/min.

Exclusion Criteria:

* prior surgical resection of the primary tumor or prior RT for lung cancer
* mixed small-cell and non-small-cell histological features
* contemporaneous immunotherapy or target therapy
* pregnancy or lactation
* physical or mental disease that could impact treatment plan
* unable to understand the trial, or could not follow the process
* to refuse the sign the informed consent.
* no history of previous malignancy in the past 5 years (except non-melanomatous skin or in situ servix carcinoma)
* be allergic to any known protocol in this trail
* be enrolled in other clinical trial in past 30days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 years
  from the starting date of treatment until the date of death from any cause

SECONDARY OUTCOMES:
Local Progression Free Survival | 5 years
  from the starting date of treatment until the date of local disease progression
Metastasis Free Survival | 5 years
  from the staring date of treatment until the date of distant metastasis
health related quality of life | from baseline, immediately after radiotherapy and an average of 3 months up to 24 months. Then through study completion, an average of 6 months.From date of randomization until the date of death from any cause, assessed up to 120 months.
  assessed from completed questionnaires. Assessments using Physicians Global Assessment to measure quality of life.
acute and late toxicity | from baseline, immediately after radiotherapy and an average of 1 week up to 12 weeks, an average of 3 months up to 24 months. Up to 120 weeks.
  acute toxicity (defined as toxicity occurring between the start of treatment and up to 3 months after completion of treatment, and assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events [version 5.0]), late toxicity (more than 3 months after completion of treatment, and assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events [version 5.0])

CONTACTS AND LOCATIONS:
Overall Officials: Anhui Shi, Doctor, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Derived] Yu J, Jiang L, Zhao L, Yang X, Wang X, Yang D, Zhuo M, Chen H, Huang W, Zhu Z, Zhang M, Song Y, Li Q, Ma Z, Wang Q, Qu Y, Yu R, Yu H, Zhao J, Shi A; Trial Management Group. High-dose hyperfractionated simultaneous integrated boost radiotherapy versus standard-dose radiotherapy for limited-stage small-cell lung cancer in China: a multicentre, open-label, randomised, phase 3 trial. Lancet Respir Med. 2024 Oct;12(10):799-809. doi: 10.1016/S2213-2600(24)00189-9. Epub 2024 Aug 12. PMID 39146944